CLINICAL TRIAL: NCT02121756
Title: A Phase I/II Pilot Study of Dipyridamole as a Modulator of Immune Activation and Systemic Inflammation in HIV-1-Infected Subjects on Antiretroviral Therapy- DAIDS-ES ID 11987
Brief Title: Dipyridamole for Immune Activation in HIV
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sharon Riddler (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Sharon Riddler, Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAIDS-ES ID 11987; U01AI110410 (NIH)
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Results first posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: HIV Infection
Keywords: Dipyridamole; HIV; Immune Markers; Immune Activation; Inflammation
MeSH Terms: conditions — HIV Infections; Inflammation | interventions — Dipyridamole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dipyridamole (Experimental): ARM A: Dipyridamole 100 mg four (4) times daily for 24 weeks from Baseline to Week 24
  Interventions: Drug: Dipyridamole
- Placebo then Dipyridamole (Active Comparator): ARM B: Placebo for Dipyridamole four (4) times daily for 12 weeks from Baseline to Week 12 followed by Dipyridamole 100mg four (4) times daily for 12 weeks from Week 12 to Week 24
  Interventions: Drug: Placebo, then Dipyridamole

INTERVENTIONS:
Drug: Dipyridamole — Dipyridamole 100 mg four (4) times daily for 24 weeks from Baseline to Week 24
  Other Names: Permole®; Persantine®
  Arms: Dipyridamole
Drug: Placebo, then Dipyridamole — Placebo for Dipyridamole four (4) times daily for 12 weeks from Baseline to Week 12 followed by Dipyridamole 100mg four (4) times daily for 12 weeks from Week 12 to Week 24
  Other Names: Permole®; Persantine®
  Arms: Placebo then Dipyridamole

SUMMARY:
The purpose of this study is to determine if Dipyridamole (DP) will decrease inflammation in HIV-1-infected individuals who are already on antiretroviral treatment and have a low viral load.

DETAILED DESCRIPTION:
Background:

* Since HIV-infected individuals started taking anti-HIV medications, illnesses from AIDS have decreased, but other serious diseases have increased. Researchers think this may be caused by an increase in activity of the immune system that fights infection, leading to inflammation. Inflammation is a normal body reaction to any infection. However, if inflammation lasts a long time, like in HIV infection, it may lead to complications such as heart disease, cancer, liver disease, lung disease, and problems with thinking. Many HIV researchers are studying the harmful effects of this prolonged immune system activity and inflammation and possible ways to prevent these complications.
* A drug called dipyridamole is approved by the Food and Drug Administration (FDA) under the trade name Persantine® for use with other drugs to reduce the risk of blood clots after heart valve replacement. Laboratory studies have shown that dipyridamole also lowers the level of immune system activity and inflammation measured in the blood.

Objectives:

* To see how dipyridamole affects blood and lung tests to measure immune system activity and inflammation and to look at the safety and tolerability of dipyridamole in people infected with HIV. This use of dipyridamole is investigational, or not approved by the FDA; however, the dose to be used in this study, 100mg four times a day, is the dose approved by the FDA.

Eligibility:

* Individuals 18 years of age and older who have HIV infection and are taking medications to treat it, and have a low viral load (HIV-1 RNA <50 copies/mL) for a minimum of 12 months.

Design:

* Participants will be screened with a physical exam, blood test, and medical history. Women of reproductive age will also receive a pregnancy test.
* Participants will take either Dipyridamole or a placebo for 12 weeks. Then they will take Dipyridamole for 12 weeks.
* During the study, participants will have frequent blood and urine tests. Dipyridamole drug levels, and liver and kidney function tests will be performed. HIV viral load (the amount of virus in the blood) will also be studied.
* Participants will have a final follow-up visit after an additional 4 weeks.
* Four brachial artery ultrasound images will be taken.
* Four pre- and post-bronchodilator spirometry tests will be performed by participants enrolled under Version 2.0: after each pre-test spirometry, participants will be asked to inhale 4 puffs of albuterol, and then to repeat the spirometry for post-testing.
* Participants will receive rectal swabs at screening, and four flexible sigmoidoscopies with rectal biopsies of the sigmoid colon throughout the study. These studies of the lower colon and samples of the rectum will be used to explore the effects of Dipyridamole. Participants can, however, opt out of all rectal procedures.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.
* On ART for at least 12 months prior to study entry with a regimen that includes three or more antiretroviral medications. More information on this criterion is available in the protocol.
* Plasma HIV-1 RNA <50 copies/mL by any standard clinical assay at screening and for a minimum of 12 months prior to entry, confirmed by at least 2 measurements prior to study entry, one of which must be at least 48 weeks prior to study entry and one of which must be 61 days and 48 weeks prior to study entry. All plasma HIV-1 RNA measurements in the 12 months prior to study entry must be <50 copies/mL (with the exception that a single detectable measurement of ≤ 200 copies/mL is permitted if the RNA levels immediately before and after are <50 copies/mL).
* Stable ART regimen for at least 8 weeks prior to study entry and no plans to change ART regimen for at least 6 months following study entry.
* Ability and willingness to provide informed consent.
* In the opinion of the investigator, no medical, mental health or other condition that precludes participation.
* Laboratory values obtained within 60 days prior to entry.

  * Hemoglobin ≥10.0 g/dL
  * Platelet count ≥100,000/mm3
  * INR ≤ 1.5 (for rectal tissue subset only)
  * PTT <2x ULN (for rectal tissue subset only)
  * AST and ALT < 2.5 x upper limit of normal (ULN)
  * Total bilirubin < 2.5 x ULN (except if hyperbilirubinemia is secondary to atazanavir).
  * Creatinine ≤ 1.5 x ULN
  * Hepatitis B surface antigen negative
  * Hepatitis C antibody negative (note: subject with HCV Ab positive is eligible if Hepatitis C RNA PCR (viral load) is undetectable)
* For females of reproductive potential, negative serum or urine pregnancy test at screening and within 72 hours prior to study entry. Females of reproductive potential include women who have not been post-menopausal for at least 24 consecutive months, (i.e., who have had menses within the preceding 24 months, or women who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy).
* Females of reproductive potential who are participating in sexual activity that could lead to pregnancy must agree to use one method of acceptable contraception while receiving protocol-specified treatment and for 4 weeks after stopping the treatment. These methods include condoms (male or female) with or without a spermicidal agent; diaphragm or cervical cap with spermicide; intrauterine device (IUD); and hormone-based contraceptive.
* Females not of reproductive potential (girls who have not reached menarche, women who have been post-menopausal for at least 24 consecutive months, or women who have undergone surgical sterilization, e.g., hysterectomy, bilateral oophorectomy, or bilateral tubal ligation or salpingectomy) are eligible without requiring the use of a contraceptive. Self- report is acceptable documentation of sterilization, other contraceptive methods, and menopause.
* Rectal Tissue Subset only: Willing to abstain from receptive anal intercourse and practices involving insertion of anything in the rectum (drug, enema, penis, or sex toy) for 72 hours prior to rectal biopsy and for 7 days post-biopsy to minimize risk of bleeding complications.

Exclusion Criteria:

* Pregnancy or breast-feeding.
* Known allergy/sensitivity or any hypersensitivity to components of study drug(s) or their formulation.
* Known cardiovascular disease (history of MI, coronary artery bypass graft surgery, percutaneous coronary intervention, stroke, transient ischemic attack, peripheral arterial disease with ABI <0.9 or claudication).
* Uncontrolled type II diabetes mellitus.
* Known chronic inflammatory conditions such as, but not limited to, rheumatoid arthritis, systemic lupus erythematosus, sarcoidosis, inflammatory bowel disease (i.e., Crohn's disease or ulcerative colitis), chronic pancreatitis, or autoimmune hepatitis, myositis, or myopathy.
* History of asthma requiring medical treatment within 2 years prior to study entry with the exception of the use of albuterol inhaler for mild intermittent asthma.
* Serious illness requiring systemic treatment and/or hospitalization within 14 days prior to entry.
* Use of any of the following medications for more than 3 consecutive days within the 60 days prior to study entry:

  * Immunosuppressives (e.g., azathioprine, corticosteroids [physiologic replacement doses are allowed], cyclosporine, mycophenolate, NSAIDs (nonsteroidal anti-inflammatory drugs), sirolimus, sulfasalazine, tacrolimus)
  * Immune modulators (e.g., cytokines [e.g., IL-2], granulocyte colony stimulating factor, growth hormone, tumor necrosis factor antagonists, thalidomide)
  * Antineoplastic agents
  * Anticoagulants (e.g., warfarin and heparin)
  * Anti-platelet drugs (e.g., clopidogrel and aspirin)
* Vaccinations within 1 week prior to the pre-entry or study entry visits. Routine standard of care vaccinations including hepatitis A and/or B, influenza, pneumococcal, and tetanus are permitted if administered at least 7 days before pre-entry and entry evaluations.
* Participation on any HIV immunotherapy or therapeutic vaccination trials within 6 months prior to study entry.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Use of investigational therapies within 30 days prior to study entry.
* Rectal Tissue Subset only:

  * Abnormalities of the colorectal mucosa or significant colorectal symptom(s), which in the opinion of the study investigator represent a contraindication to biopsy (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, and presence of symptomatic external hemorrhoids.
  * NOTE: Abnormalities of the colorectal mucosa will be assessed at the time of the enrollment flexible sigmoidoscopy. If no significant colorectal abnormalities or symptoms are present then the participant will undergo the enrollment procedures. If abnormalities are present then no biopsies will be performed and the participant will not be enrolled into the rectal tissue subset but will continue participation in the main study.
  * Active untreated gonorrhea, or chlamydia infection within 30 days prior to study entry (subjects diagnosed with rectal gonorrhea or chlamydia infection at screening may be treated during the screening period provided the treatment is at least 30 days prior to entry).
* Exclusions for spirometry testing (for participants enrolled under Version 2.0) Participants will not undergo pre- and post-bronchodilator spirometry if they have any of the following: - Abdominal or cataract surgery within 3 months.

  * Myocardial infarction or stroke within the past 3 months.
  * Acute onset of shortness of breath, cough, fever or heart condition such as tachycardia, angina or arrhythmias with 4 weeks prior to enrollment.
  * Increasing respiratory symptoms or febrile (temperature >100.4°F [38°C]) within 4 weeks of study entry.
  * Uncontrolled hypertension defined as systolic > 160 mm Hg or diastolic > 100 mm Hg from an average of two or more readings. Participant with controlled hypertension may undergo spirometry.
  * Prior history of adverse reaction to albuterol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A. Riddler, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Pitt Treatment Evaluation Unit / University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ARM A: Dipyridamole for 24 Weeks: Dipyridamole 100 mg four (4) times daily for 24 weeks from Baseline to Week 24
- ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks: Placebo for Dipyridamole four (4) times daily for 12 weeks from Baseline to Week 12 followed by Dipyridamole 100mg four (4) times daily for 12 weeks from Week 12 to Week 24
Period: Overall Study
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Started | 21 | 19
Completed | 15 | 17
Not Completed | 6 | 2
Not completed — Adverse Event | 3 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: 40 HIV-1-infected, ART-treated adults 18 years of age and older with HIV-1 RNA less than 50 copies/mL were enrolled and randomized. Of these 40 participants, 35 participants were included in the as-treated (AT) analysis (17 Dipyridamole, 18 placebo).
Groups:
- ARM B: Placebo for 12 Weeks, Then Dipyridamole for 12 Weeks: Placebo for Dipyridamole four (4) times daily for 12 weeks from Baseline to Week 12 followed by Dipyridamole 100mg four (4) times daily for 12 weeks from Week 12 to Week 24
- Total: Total of all reporting groups
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks, Then Dipyridamole for 12 Weeks | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 19 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (11.2) | 50.0 (6.9) | 49.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 20 | 15 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 15 | 13 | 28
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 19 | 40
sCD14 plasma levels [Median (Inter-Quartile Range); unit: pg/ml] — Population: 35 participants were included in the as-treated (AT) analysis (17 Dipyridamole, 18 placebo); 4 Dipyridamole (1 adverse event 1 protocol deviation, 2 investigator discretion) and 1 placebo (change in antiretroviral therapy) participants were excluded from the primary AT analysis.
  pg/ml
    number analyzed (Participants) | 17 | 18 | 35
    (all) | 1634000.00 [1350801.50 to 2048500.00] | 1754500.00 [1345500.00 to 2215500.00] | 1695500.00 [1345500.00 to 2134000.00]
sCD163 plasma levels [Median (Inter-Quartile Range); unit: ng/ml] — Population: 35 participants were included in the as-treated (AT) analysis (17 Dipyridamole, 18 placebo); 4 Dipyridamole (1 adverse event 1 protocol deviation, 2 investigator discretion) and 1 placebo (change in antiretroviral therapy) participants were excluded from the primary AT analysis.
  ng/ml
    number analyzed (Participants) | 17 | 18 | 35
    (all) | 478.81 [404.63 to 767.90] | 528.09 [422.27 to 738.40] | 525.49 [404.63 to 767.90]
IL-6 plasma levels [Median (Inter-Quartile Range); unit: pg/ml] — Population: 35 participants were included in the as-treated (AT) analysis (17 Dipyridamole, 18 placebo); 4 Dipyridamole (1 adverse event 1 protocol deviation, 2 investigator discretion) and 1 placebo (change in antiretroviral therapy) participants were excluded from the primary AT analysis.
  pg/ml
    number analyzed (Participants) | 17 | 18 | 35
    (all) | 1.30 [0.83 to 2.00] | 1.77 [1.08 to 3.20] | 1.48 [1.06 to 2.68]

OUTCOME MEASURES:

1. Primary Outcome: Monocyte and Macrophage Activation Assessed as Change in Plasma Levels of sCD14 From Baseline to Week 12
Description: Change in plasma levels of sCD14 from baseline to week 12
Time Frame: Baseline to week 12
Population: 35 participants were included in the as-treated (AT) analysis (17 Dipyridamole, 18 placebo); 4 Dipyridamole (1 adverse event 1 protocol deviation, 2 investigator discretion) and 1 placebo (change in antiretroviral therapy) participants were excluded from the primary AT analysis.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- ARM A: Dipyridamole for 24 Weeks: ARM A: Dipyridamole 100 mg four (4) times daily for 24 weeks from Baseline to Week 24
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 17 | 18
pg/ml | 244500.00 [-318792.00 to 479000.00] | -58250.00 [-572567.50 to 287500.00]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other — The sCD14 is measured in pg/ml and the median change is shown in pg/ml. the linear regression for the between arm comparison of baseline to week 12 change was performed using log10 transformed plasma sCD14; p = 0.8220, Regression, Linear

2. Primary Outcome: Monocyte and Macrophage Activation Assessed as Change in Plasma Levels of sCD163 From Baseline to Week 12
Description: Change in Plasma levels of sCD163 from baseline to week 12
Time Frame: baseline to week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 17 | 18
ng/ml | -6.19 [-78.04 to 25.93] | 5.42 [-38.33 to 88.33]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other — The sCD163 is measured in ng/ml and the median change is shown in ng/ml. the linear regression for the between arm comparison of baseline to week 12 change was performed using log10 transformed plasma sCD163; p = 0.0869, Regression, Linear

3. Primary Outcome: Systemic Inflammation Assessed as Change in IL-6 Plasma Levels From Baseline to Week 12
Description: Change in Plasma levels of IL-6 from baseline to week 12
Time Frame: baseline to week 12
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 17 | 18
pg/ml | -0.02 [-0.36 to 0.86] | -0.07 [-0.59 to 0.88]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other — The IL-6 is measured in pg/ml and the median change is shown in pg/ml. the linear regression for the between arm comparison of baseline to week 12 change was performed using log10 transformed plasma IL-6; p = 0.5027, Regression, Linear

4. Secondary Outcome: Immune System Activation as Measured by the Proportion of CD8+ T Cells Co-expressing CD69 and CD25 After 12 Weeks of Dipyridamole Treatment Compared to Placebo
Description: To compare changes in the level of T cell immune activation as measured by the proportion of CD8+ T cells co-expressing CD69 and CD25 after 12 weeks of Dipyridamole treatment to placebo.
Time Frame: Baseline to week 12
Population: Per protocol, participants randomized to placebo were crossed over to DP after week 12.
Measure: Median (Inter-Quartile Range); unit: proportion of CD8+ T cells
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 17 | 18
proportion of CD8+ T cells | -0.05 [-0.15 to 0.00] | 0.00 [-0.05 to 0.05]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other; p = 0.4548, Mixed Models Analysis

5. Secondary Outcome: Safety and Tolerability of Dipyridamole Assessed as the Number of Participants With Grade 2 or Higher Adverse Events or Treatment Discontinuations
Description: Grade 2 or higher adverse events and treatment discontinuations
Time Frame: First 12 weeks of dipyridamole treatment
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 21 | 19
Participants
  Grade 2 adverse events | 12 | 10
  Grade 3 adverse events | 2 | 1
  Treatment discontinuations | 4 | 0
  No Grade 2 or 3 AEs or treatment discontinuations | 3 | 8

6. Secondary Outcome: Immune System Activation Assessed as the Change in the Proportion of Cycling CD4+ T Cells as Measured by Ki-67 Expression at Baseline and After Treatment With Dipyridamole
Description: To assess whether Dipyridamole reduces the proportion of cycling CD4+ T cells as measured by Ki-67 expression at baseline and after treatment with Dipyridamole.
Time Frame: Baseline to week 12
Population: Per protocol, participants randomized to placebo were crossed over to DP after week 12.
Measure: Median (Inter-Quartile Range); unit: proportion of cycling CD4+ T Cells
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 17 | 18
proportion of cycling CD4+ T Cells | -0.15 [-0.30 to -0.05] | -0.05 [-0.20 to 0.05]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other; p = 0.7556, Mixed Models Analysis

7. Secondary Outcome: Immune System Activation as Measured by the Proportion of CD4+ T Cells Co-expressing HLA-DR and CD38 After 12 Weeks of Dipyridamole Treatment Compared to Placebo
Description: To compare changes in the level of T cell immune activation as measured by the proportion of CD4+ T cells co-expressing HLA-DR and CD38 after 12 weeks of DP treatment to placebo.
Time Frame: Baseline to week 12
Population: Per protocol, participants randomized to placebo were crossed over to DP after week 12.
Measure: Median (Inter-Quartile Range); unit: proportion of CD4+ T cells
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 17 | 18
proportion of CD4+ T cells | -0.25 [-0.70 to 0.00] | 0.10 [-0.65 to 0.55]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other; p = 0.2075, Mixed Models Analysis

8. Secondary Outcome: Immune System Activation as Measured by the Proportion of CD8+ T Cells Co-expressing HLA-DR and CD38 After 12 Weeks of Dipyridamole Treatment Compared to Placebo
Description: To compare changes in the level of T cell immune activation as measured by the proportion of CD8+ T cells co-expressing HLA-DR and CD38 after 12 weeks of Dipyridamole treatment to placebo.
Time Frame: Baseline to week 12
Population: Per protocol, participants randomized to placebo were crossed over to Dipyridamole after week 12.
Measure: Median (Inter-Quartile Range); unit: proportion of CD8+ T cells
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 17 | 18
proportion of CD8+ T cells | -0.85 [-2.35 to 0.30] | 0.25 [-0.40 to 1.80]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other; p = 0.0315, Mixed Models Analysis

9. Secondary Outcome: Immune System Activation Assessed by the Proportion of CD4+ T Cells Co-expressing CD69 and CD25 After 12 Weeks of Dipyridamole Treatment to Placebo
Description: To compare changes in the level of T cell immune activation as measured by the proportion of CD4+ T cells co-expressing CD69 and CD25 after 12 weeks of Dipyridamole treatment to placebo.
Time Frame: Baseline to week 12
Population: Per protocol, participants randomized to placebo were crossed over to Dipyridamole after week 12.
Measure: Median (Inter-Quartile Range); unit: proportion of CD4+ T cells
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 17 | 18
proportion of CD4+ T cells | 0.00 [-0.20 to 0.20] | 0.00 [-0.05 to 0.10]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other; p = 0.7376, Mixed Models Analysis

10. Secondary Outcome: Cellular Immune Activation: Change in the Proportion of Cycling CD8+ T Cells
Description: To assess whether Dipyridamole reduces the proportion of cycling CD8+ T cells as measured by Ki-67 expression at baseline and after treatment with Dipyridamole.
Time Frame: Baseline to week 12
Population: Per protocol, participants randomized to placebo were crossed over to Dipyridamole after week 12.
Measure: Median (Inter-Quartile Range); unit: proportion of cycling CD8+ T Cells
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 17 | 18
proportion of cycling CD8+ T Cells | -0.20 [-0.50 to 0.05] | 0.05 [-0.20 to 0.20]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other; p = 0.2343, Mixed Models Analysis

11. Secondary Outcome: Systemic Inflammatory Biomarkers: Change in the Levels of sTNFαR
Description: To compare changes in the levels of sTNFαR after 12 weeks of dipyridamole treatment to placebo
Time Frame: Baseline to week 12
Population: Per protocol, participants randomized to placebo were crossed over to Dipyridamole after week 12.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 16 | 18
pg/ml | -84.61 [-287.58 to 492.48] | 34.26 [-284.50 to 495.36]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other; p = 0.7598, Mixed Models Analysis

12. Secondary Outcome: Systemic Inflammatory Biomarkers: Change in the Levels of TNFα
Description: To compare changes in the levels of TNFα after 12 weeks of dipyridamole treatment to placebo
Time Frame: Baseline to week 12
Population: Per protocol, participants randomized to placebo were crossed over to Dipyridamole after week 12.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 16 | 18
pg/ml | -152.31 [-1430.45 to 1874.43] | 123.88 [-625.73 to 963.73]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other; p = 0.9830, Mixed Models Analysis

13. Secondary Outcome: Systemic Inflammatory Biomarkers: Change in the Levels of hsCRP
Description: To compare changes in the levels of hsCRP after 12 weeks of dipyridamole treatment to placebo
Time Frame: Baseline to week 12
Population: Per protocol, participants randomized to placebo were crossed over to Dipyridamole after week 12.
Measure: Median (Inter-Quartile Range); unit: ng/dl
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 17 | 18
ng/dl | -233.57 [-699.19 to 970.26] | -750.35 [-4385.43 to 201.94]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other; p = 0.3317, Mixed Models Analysis

14. Secondary Outcome: Coagulation Biomarkers: Change in the Levels of D-dimer
Description: To compare changes in the levels of D-dimer after 12 weeks of dipyridamole treatment to placebo
Time Frame: Baseline to week 12
Population: Per protocol, participants randomized to placebo were crossed over to Dipyridamole after week 12.
Measure: Median (Inter-Quartile Range); unit: mcg/ml
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 17 | 18
mcg/ml | 45.86 [-7.88 to 142.07] | 36.35 [-15.44 to 187.07]
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other; p = 0.6121, Mixed Models Analysis

15. Secondary Outcome: Changes in Brachial Artery Flow-mediated Dilation (FMD)
Description: To compare % change at tmax in brachial artery flow-mediated dilation (FMD) after 12 weeks of dipyridamole treatment to placebo
Time Frame: Baseline to week 12
Population: Per protocol, participants randomized to placebo were crossed over to DP after week 12.
Measure: Mean (Standard Deviation); unit: percentage change at tmax
Arm/Group | ARM A: Dipyridamole for 24 Weeks | ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks
Number analyzed (Participants) | 14 | 17
percentage change at tmax | 0.1 (5.2) | -1.1 (4.8)
Statistical Analysis 1: Comparison: ARM A: Dipyridamole for 24 Weeks vs ARM B: Placebo for 12 Weeks Then Dipyridamole for 12 Weeks; Test type: Other; p = 0.5620, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Baseline to Week 24
Groups:
- ARM A: Dipyridamole for 24 Weeks From Baseline to Week 24: ARM A: Summary of Adverse Events for all participants randomized to receive Dipyridamole 100 mg four (4) times daily for 24 weeks from Baseline to Week 24
- ARM B: Placebo for 12 Weeks From Baseline to Week 12: ARM B: Summary of Adverse Events for all participants randomized to receive Placebo for Dipyridamole four (4) times daily for 12 weeks from Baseline to Week 12
- ARM B: Dipyridamole for 12 Weeks From Week 12 to Week 24: ARM B: Summary of Adverse Events for all participants randomized to receive Dipyridamole 100mg four (4) times daily for 12 weeks from Week 12 to Week 24
Arm/Group | ARM A: Dipyridamole for 24 Weeks From Baseline to Week 24 | ARM B: Placebo for 12 Weeks From Baseline to Week 12 | ARM B: Dipyridamole for 12 Weeks From Week 12 to Week 24
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 20/21 | 14/19 | 12/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A: Dipyridamole for 24 Weeks From Baseline to Week 24 (N=21) | ARM B: Placebo for 12 Weeks From Baseline to Week 12 (N=19) | ARM B: Dipyridamole for 12 Weeks From Week 12 to Week 24 (N=19)
gastrointestinal (Gastrointestinal disorders) | 13 (49) | 8 (16) | 5 (18)
Neurologic (Nervous system disorders) | 13 (28) | 5 (6) | 6 (11)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 8 (13) | 2 (3) | 4 (4)
cardiovascular (Cardiac disorders) | 6 (12) | 1 (1) | 3 (3)
respiratory (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 1 (1) | 5 (5)
endocrine/metabolic (Endocrine disorders) | 3 (4) | 0 (0) | 1 (1)
chemistries (Investigations) | 2 (3) | 2 (2) | 0 (0)
systemic (General disorders) | 4 (7) | 2 (2) | 2 (3)
genitourinary (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
dermatologic (Skin and subcutaneous tissue disorders) | 4 (6) | 2 (2) | 1 (1)
hematologic (Investigations) | 2 (2) | 0 (0) | 0 (0)
infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
ocular/visual (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
psychological/emotional (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-02-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT02121756/Prot_SAP_000.pdf
  • Informed Consent Form (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/56/NCT02121756/ICF_001.pdf